CLINICAL TRIAL: NCT02439528
Title: Genetics of the Combined Pulmonary Fibrosis and Emphysema Syndrome
Acronym: GENES-SEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2013.819
Record Dates: First submitted 2014-08-29; First posted 2015-05-08 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Combined Pulmonary Fibrosis and Emphysema Syndrome; Pulmonary Fibrosis; Emphysema; Healthy Subjects
Keywords: pulmonary fibrosis; syndrome; genetic; emphysema
MeSH Terms: conditions — Pulmonary Fibrosis; Emphysema; Syndrome | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Combined pulmonary fibrosis and emphysema syndrome (Other): Genetic analysis on patients with combined pulmonary fibrosis and emphysema syndrome.
  Interventions: Genetic: Genetic analysis
- Pulmonary fibrosis (Other): Genetic analysis on patients with pulmonary fibrosis.
  Interventions: Genetic: Genetic analysis
- Emphysema (Other): Genetic analysis on patients with emphysema.
  Interventions: Genetic: Genetic analysis
- Healthy subject (Other): Genetic analysis on healthy subject.
  Interventions: Genetic: Genetic analysis

INTERVENTIONS:
Genetic: Genetic analysis — One part of these patients is already included in a cohort: for them the blood sample will be centralized and then analyzed.
  The other part of these patients will be recruited during the study: for them intervention will be blood samples for further genetic analysis.

SUMMARY:
The combined pulmonary fibrosis and emphysema syndrome (CPFE) individualized by our group in 2005 is characterized by an often severe dyspnea, almost exclusive male predominance, and often major, profound impairment of gas exchange contrasting with preserved lung volumes and absence of airflow obstruction, and a high risk of pre-capillary pulmonary hypertension responsible for increased mortality. Almost all patients are smokers or ex-smokers. There are some arguments in favor of genetic abnormalities in this syndrome of unknown etiology (other than smoking) including short telomeres and mutations in the telomerase complex genes. There are also emphysematous lesions, in patients with familial pulmonary fibrosis, with mutations in the SFTPC gene (surfactant protein C), and reported cases of CPFE syndrome with SFTPC mutation. No large genetic studies have been conducted to date in the CPFE syndrome. Our main hypothesis is that the proportion of subjects with short telomeres is higher among patients with CPFE syndrome than in subjects of similar age with idiopathic pulmonary fibrosis but without emphysema. It has previously been shown that mutations in the telomerase TERT or TERC genes are mostly found in people whose telomeres are abnormally short. The investigators propose to use that test to identify patients most likely carrying a mutation, and to seek, among them, the mutations in the TERT or TERC telomerase genes. The objective of the study is to compare the proportion of patients with short telomeres in the group of patients with CPFE syndrome to that of other patients (with idiopathic pulmonary fibrosis without emphysema, or with emphysema without fibrosis).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years old.
* Patient with Idiopathic Pulmonary Fibrosis Or
* Patient with emphysema Or
* Patient with combined pulmonary fibrosis and emphysema syndrome Or
* Patient reporting no chronic lung disease

Exclusion Criteria:

* Other causes of interstitial lung disease or context:

  * Connective
  * Pneumonia drug
  * Pneumoconiosis
  * Sarcoidosis
  * histiocytosis, lymphangioleiomyomatosis, etc.
* Refusal to participate in the study or to sign the consent
* Inability to give informed about the information
* Woman breastfeeding or pregnant
* No coverage for Social Security
* Deprivation of Civil Rights

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
Telomere length | At inclusion
  The primary endpoint is the percentage of patients with telomere length less than the 10th percentile of the age range for each type of patient

SECONDARY OUTCOMES:
Mutation of the telomerase complex genes evaluated by gene sequencing. | At inclusion
  Frequency of the telomerase complex mutations measured by the percentage of patients having at least one mutation of the complex.
Mutations in the gene encoding the SFTPC evaluated by gene sequencing | At inclusion
  Frequency of mutations in the gene encoding the SFTPC surfactant protein C measured by the percentage of patients having at least one mutation of the complex
Patients characteristics evaluated by clinical examination | At inclusion
  Comparison of each type of patients with controls
Genetic profile evaluated by gene sequencing. | At inclusion
  Description of the mutations found, relations with the phenotype
Total mortality evaluated by phone call contact | 6 months
  6 months after inclusion, patients will be contacted to know their clinical status.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent COTTIN, MD, Principal Investigator — Hospices Civils de Lyon
Locations (3):
- France (3):
  - Hôpital pneumologique et cardiovasculaire Louis Pradel, HCL, Bron
  - Hôpital Albert Michallon, CHU de Grenoble, Grenoble
  - Hôpital Nord, CHU de Saint-Etienne, Saint-Etienne